CLINICAL TRIAL: NCT05992480
Title: An Open-Label, Case-Control Study to Compare the Anamnestic Response to the Recombinant Vesicular Stomatitis Delta Glycoprotein Zaire Ebola Virus (ZEBOV) Glycoprotein (rVSVDG-ZEBOV-GP) Ebola Virus Vaccine Among Ebola Virus Disease Survivors to the Primary Immune Response Among Naïve Age and Sex-Matched Controls
Brief Title: REVIVE (Response to the Ebola Virus Vaccine)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Kenema Government Hospital (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-970
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Ebola Virus Disease
Keywords: Vaccine; Ebola; Sierra Leone; Ebola survivor
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Intervention Model Description: 1:1 survivor to control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ebola Virus Disease (EVD) survivors (Experimental): Participants with a history of admission and discharge from an Ebola Treatment Unit as registered by the Sierra Leone Association of Ebola Survivors (SLAES), and Anti-EBOV GP IgG positive by ELISA at the time of screening.
  Interventions: Biological: rVSVDG-ZEBOV-GP Ebola Virus Vaccine (ERVEBO)
- Community control (Active Comparator): Age- and sex-matched controls who are Anti-EBOV GP IgG negative by ELISA at the time of screening.
  Interventions: Biological: rVSVDG-ZEBOV-GP Ebola Virus Vaccine (ERVEBO)

INTERVENTIONS:
Biological: rVSVDG-ZEBOV-GP Ebola Virus Vaccine (ERVEBO) — It is an Ebola virus vaccine

SUMMARY:
This study is a vaccine-related clinical trial which will be conducted by our study team at Kenema Government Hospital (KGH)'s Viral Hemorrhagic Fever Program in collaboration with Tulane University School of Medicine. This study is funded by Merck & Co., the developers of ERVEBO®. This investigational medicinal product (IMP) was successful in Sierra Leone through the Sierra Leone Trial to Introduce a Vaccine against Ebola (STRIVE) working with the College of Medical and Allied Health Services (COMAHS) at the University of Sierra Leone. ERVEBO® was also successfully tested in Liberia and the Republic of Guinea. These successful trials led to the United States Food and Drug Administration (USFDA) approval of ERVEBO®, as well as approval for therapeutic use in the Democratic Republic of the Congo, Burundi, Ghana, and Zambia.

This particular vaccination study will focus on the anamnestic response to the ERVEBO® vaccine, (full name - rVSVDG-ZEBOV-GP Ebola Virus Vaccine). The original clinical trials conducted excluded Ebola Virus Disease (EVD) survivors from participating. However, with ongoing research, there is evidence of waning immune response and even recurrent infections in EVD survivors.

DETAILED DESCRIPTION:
Ebola virus (EBOV; also known as Zaire ebolavirus, family Filoviridae) is among the most virulent infectious agents known, producing sporadic outbreaks of severe and highly lethal hemorrhagic fever in humans and nonhuman primates (NHPs). The West African Ebola Virus Disease (EVD) Outbreak of 2013 to 2016, which predominantly affected Sierra Leone, Liberia, and Guinea, resulted in 28,601 confirmed cases and 11,308 fatalities.

Multiple reports in the literature of recurrent infections among EVD survivors now exist. Some of these recurrent infections have also resulted in transmission to close contacts of these survivors. In December 2019, the U.S. Food and Drug Administration approved the recombinant Vasicular Stomatitis Virus delta-G (rVSVDG) Zaire Ebolavirus (ZEBOV) Glycoprotein (GP) (rVSVDG-ZEBOV-GP) Ebola vaccine (ERVEBO®; Merck) for use in people 18 years and older. The current literature and data on EBOV antibody levels in survivors suggest that while the humoral immune response to EBOV after natural infections wanes over weeks to months, the response to a single dose of rVSVDG-ZEBOV-GP vaccine is stable over at least two years.

In this pilot study, the investigators hypothesize that vaccination of EVD survivors with rVSVDG-ZEBOV-GP will result in a non-inferior immune response compared to vaccination of non-exposed age- and sex-matched individuals. This study will be an open-label, case-control study of the safety and immunogenicity of the rVSVDG-ZEBOV-GP vaccine comparing EVD survivors and EBOV-naïve community members in Sierra Leone. A total of 40 participants will be recruited and divided 1:1 into EVD survivors (cases) and EBOV-naïve age- and sex-matched community members (controls). Following a two week screening period, participants will be followed for six months post-vaccination.

Subject Population

Twenty EVD survivors and twenty age and sex-matched controls with no clinical history or immunologic evidence of prior EBOV infection will be enrolled. All participants will be citizens of Sierra Leone. In accordance with the currently approved use of the rVSVDG-ZEBOV-GP vaccine in Sierra Leone, all participants will be 18 years or older and pregnant and lactating females will be excluded.

While there is currently an effort to vaccinate all healthcare workers in Sierra Leone, EVD survivors are excluded in the current vaccine roll-out. The investigators plan to recruit EVD survivors including healthcare workers thus enhancing access to the vaccine for this population. All participants will be of African descent. The investigators plan to enroll an equal number of males and females.

ELIGIBILITY:
Inclusion Criteria:

* EVD survivors

  * History of admission and discharge from an Ebola Treatment Unit as registered by the Sierra Leone Association of Ebola Survivors (SLAES).
  * Anti-EBOV GP IgG positive by ELISA at the time of screening.
  * ≥18 years of age.
  * >45.5 kg (100lbs).
  * Willingness to provide informed, written consent.
  * Willingness to undergo all study procedures including rVSVDG-ZEBOV-GP vaccination and multiple blood collections over a period of six months.
* Age- and sex-matched controls

  * Anti-EBOV GP IgG negative by ELISA at the time of screening.
  * ≥18 years of age.
  * Willingness to provide informed consent.
  * Willingness to undergo all study procedures including rVSVDG-ZEBOV-GP vaccination and multiple blood collections over a period of six months.

Exclusion Criteria:

* Have received the rVSVDG-ZEBOV-GP vaccine.
* Currently participating in another clinical trial involving a vaccine.
* Received a live vaccine within four weeks of screening.
* <18 years of age.
* Weight <45.5kg (or 100 lbs).
* Refusal to provide informed, written consent.
* Prisoners of other institutionalized individuals.
* Research study staff and their immediate family members.
* Inability to participate in research activities.
* Pregnant and lactating females.
* Known immunocompromised status.
* Known allergy to vaccine components.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assess the immunogenicity and durability of rVSVDG-ZEBOV-GP among EVD survivors compared with unexposed age- and sex-matched controls at six months post-vaccination | 6 months
  Serum samples will be tested for the presence of anti-EBOV GP immunoglobulin G (IgG) and anti-EBOV Viral Protein 40 (VP40) IgG using ELISA plates produced by Zalgen Labs, LLC and run according to the manufacturer's instructions.
Assess the incidence of adverse events after vaccination with rVSVDG-ZEBOV-GP among EVD survivors compared with unexposed age- and sex-matched controls | 6 months
  The investigators will assess the following adverse events at all post-vaccination follow-up time points: arthralgia, diarrhea, fatigue, fever, headache, induration, injection site pain, muscle pain, myalgia, and vomiting. Follow up visits will occur on days 1, 3, 7, 14, 28, 90 and 180 post vaccination.

SECONDARY OUTCOMES:
Assess the durability of neutralizing antibody titers after immunization with rVSVDG-ZEBOV-GP among EVD survivors compared with unexposed age- and sex-matched controls at six months post-vaccination | 6 months
  The investigators will use Pseudovirus Neutralization Assay that has been adapted from a previously described Lassa pseudovirus to produce Ebola pseudoviruses (EBOVpp). EBOVpp are capable of a single round of replication, when used to infect a human embryonic kidney cell line which is capable of fluorescence.
Determine Fc-mediated innate effector function profiles in EVD survivors compared to both naïve vaccinees and EVD survivors vaccinated with rVSVDG-ZEBOV-GP. | 6 months
  The investigators will use a bead-based multiplexed platform to measure Fc-mediated effector functional profiles and virus specific antibodies using an established EBOV systems serology platform including: (A) monocyte/macrophage phagocytosis and activation, (B) neutrophil phagocytosis and maturation, (C) Natural Killer (NK) cell activation, and (D) complement deposition.
Assess the phenotype, function, and durability of EBOV specific T-cell responses in natural immunity (EVD survivors) and response to vaccination with rVSVDG-ZEBOV-GP in EVD survivors and naïve vaccinees | 6 months
  EBOV specific T-cells will be characterized by: (A) EBOV protein stimulation and intracellular cytokine staining, (B) magnetic bead-based assays to assess function in supernatants from stimulated cells, and (C) Two-color Interferon-Gamma and Tumor Necrosis Factor-Alpha (TNFa) Enzyme Linked Immunosorbent Spot (ELISPOT).

CONTACTS AND LOCATIONS:
Overall Officials: John Schieffelin, MD, Principal Investigator — Tulane University
Locations (1):
- Kenema Government Hospital, Kenema, Eastern Province, Sierra Leone

IPD SHARING:
Plan to Share IPD: Yes
The Principal Investigator or their designee will be the data manager with responsibility for delegating the receiving, entering, cleaning, querying, analyzing, and storing all data accrued from the study. All data will be entered in paper case record forms and transcribed by double entry into an electronic database. This includes safety data, laboratory data (both clinical and immunological) and outcome data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From preliminary interim analysis until the final report of the study, the site owns the data and it is agreed that publication will occur in a timely manner.
Access Criteria: All files and source documents will be kept confidentially in locked, fireproof safety cabinets with limited access. The Principal Investigator, co-investigators, and clinical research staff will have access to records. The investigators will permit authorized representatives of the sponsor, regulatory agencies, and monitors to examine (and when required by applicable law, to copy) clinical records for the purposes of quality assurance reviews, audits, and evaluation of the study safety and progress.